CLINICAL TRIAL: NCT06841484
Title: Clinical Outcomes of Full Robotic Instrumentation Versus Assistant Controlled Laparoscopic Instrumentatin in Robotic Distal Gastrectomy: Randomized Pilot Study
Brief Title: Comparison of Full Robotic Instrumentation and Assistant-Controlled Laparoscopic Instrumentation in Robotic Distal Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2024-0426
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Blind Randomized controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assistant-Controlled Group (Experimental): The assistant performs vascular clipping using articulating Hemolock clip appliers or Challenger® clip appliers and performs the gastrointestinal anastomosis with an Echelon stapling system.
  Interventions: Procedure: Arm I (Assistant-Controlled Laparoscopic Instrumentation)
- Full Robotic Group (Active Comparator): The surgeon performs vascular clipping using the robotic arm with Hemolock or Hemoclip appliers and performs anastomosis using a SureForm stapler.
  Interventions: Procedure: Arm II (Assistant-Controlled Laparoscopic Instrumentation)

INTERVENTIONS:
Procedure: Arm I (Assistant-Controlled Laparoscopic Instrumentation) — In this group, robotic distal gastrectomy is performed with assistant-controlled laparoscopic instrumentation. The assistant conducts vascular clipping using articulating Hemolock clip appliers (Livsmed) or Challenger® clip appliers (B.Braun). For gastrointestinal anastomosis, the assistant operates an Echelon stapling system (Johnson & Johnson) via the assistant port. The surgeon controls the robotic console for all other surgical steps. This method utilizes a hybrid approach, combining robotic precision with laparoscopic efficiency.
  Arms: Assistant-Controlled Group
Procedure: Arm II (Assistant-Controlled Laparoscopic Instrumentation) — In this group, all surgical steps, including vascular clipping and anastomosis, are performed using the robotic system. The surgeon utilizes the Da Vinci Xi system and switches robotic instruments as needed. Vascular clipping is performed with robotic Hemolock or Hemoclip appliers, and anastomosis is conducted using the SureForm robotic stapler. This fully robotic technique eliminates laparoscopic assistance and utilizes only robotic arms for the entire procedure.
  Both groups follow the same postoperative care protocols, including standardized pain management and recovery assessments.
  Arms: Full Robotic Group

SUMMARY:
This pilot study aims to provide valuable insights into the optimal surgical approach for robotic distal gastrectomy. By comparing full robotic procedures with assistant-controlled techniques, the results may guide future practice, enhancing surgical efficiency, reducing costs, and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed gastric adenocarcinoma prior to surgery.
2. Patients who have undergone a complete (R0) resection.
3. Patients with an ASA (American Society of Anesthesiologists) score of 3 or below.
4. Patients undergoing robotic radical distal gastrectomy.

Exclusion Criteria:

1. Patients under 19 years of age.
2. Patients who have received preoperative chemotherapy or radiotherapy.
3. Patients diagnosed with stage IV gastric cancer due to distant metastasis.
4. Patients diagnosed with malignancies other than gastric cancer.
5. Patients scheduled to undergo total gastrectomy.
6. Patients requiring total omentectomy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Average operative time (in minutes). | At the end of the surgery
  The primary outcome is the average operative time (in minutes) from skin incision to skin closure. This measurement will compare surgical efficiency between the assistant-controlled laparoscopic instrumentation group and the full robotic instrumentation group.

SECONDARY OUTCOMES:
Total cost of consumable surgical materials. | At the end of the surgery (up to 12 hours)
  The total cost of surgical consumables, including robotic instruments, staplers, clips, and other disposable materials used during the procedure, will be calculated from the surgical expense records.
Quality of Recovery (QoR-15) scores at 72 hours postoperatively. | 72 hours postoperatively
  The total cost of surgical consumables, including robotic instruments, staplers, clips, and other disposable materials used during the procedure, will be calculated from the surgical expense records.
Time to first flatus and bowel movement. | Up to 1 month after surgery
  The time taken for the patient to pass gas and have a bowel movement will be recorded to assess postoperative gastrointestinal recovery.
Postoperative laboratory markers (e.g., CRP, WBC). | Up to 5 days after surgery
  Inflammatory markers, including C-reactive protein (CRP) and white blood cell (WBC) counts, will be measured from blood samples to evaluate the patient's inflammatory response.
Incidence of postoperative complications. | Within 30 days postoperatively
  The incidence of postoperative complications, including infections, bleeding, anastomotic leakage, and other surgical site issues, will be recorded and classified according to the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeveranceHospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided